CLINICAL TRIAL: NCT03611504
Title: Hemospray Effectiveness and Predictors of Rebleeding in Patients With Gastrointestinal Hemorrhage: A Real-life Multicenter Cohort.
Brief Title: Hemospray in Gastrointestinal Bleeding: A Real-life Multicenter Cohort
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: University of Salamanca (Other); Hospital del Mar (Other); Puerta de Hierro University Hospital (Other); Complejo Hospitalario de Navarra (Other); Hospital de Henares (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Quirón Madrid University Hospital (Other); Hospital de Cruces (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Central de Asturias (Other); Hospital Universitario de Cabuenes (Other); Hospital Universitario Doctor Peset (Other); Hospital del Rio Hortega (Other); Hospital Universitario Madrid Sanchinarro (Other); Hospital de Aviles (Unknown); Hospital IMQ Zorrozaurre (Unknown)
Responsible Party: Principal Investigator, Enrique Rodríguez de Santiago, M.D Gastroenterologist, Hospital Universitario Ramon y Cajal
Other Study IDs: HRC-HEMOSPRAY
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Gastrointestinal Hemorrhage; Ulcer Hemorrhage; Tumor Bleeding
Keywords: Hemospray, Gastrointestinal bleeding, Gastrointestinal hemorrhage, Hemostatic powder
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hemospray® group: Patients with gastrointestinal bleeding treated with Hemospray®.
  Interventions: Device: Hemospray®

INTERVENTIONS:
Device: Hemospray® — Hemospray® application
  Other Names: Hemostatic powder

SUMMARY:
This is an observational, retrospective, analytical, and multicenter study conducted at 17 hospitals. Our research aims to assess the effectiveness of Hemospray® in patients with gastrointestinal bleeding in clinical practice. Besides, we aim to detect predictors of treatment failure defined as unsuccessful immediate hemostasis or rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastrointestinal bleeding treated with Hemospray®.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gastrointestinal bleeding treated with Hemospray®.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Hemospray® intraprocedural bleeding control | From Hemospray® first application up to the end of the endoscopic procedure. This variable should be assessed in day 1.
  It refers to the proportion (%) of patients who achieves intraprocedural hemostasis with Hemospray®. Intraprocedural bleeding control is defined as endoscopic observation of bleeding cessation after Hemospray® use.
Rebleeding rate | Date of Hemospray® application until rebleeding, assessed up to 48 months
  To describe the rebleeding rate (%) after Hemospray®. Rebleeding is defined as a new episode of hematemesis, rectorrhagia or melena; hemoglobin level decrease >2 g/dL within 48 h of the index endoscopy or direct visualization of active bleeding at the previously treated lesion at repeat endoscopy.

SECONDARY OUTCOMES:
Adverse events potentially related to Hemospray® | From Hemospray application until day +7
  Abdominal distension (Yes/no), Intestinal perforation (Yes/No). Unexpected adverse events will be also recorded and evaluated.
Mortality | From Hemospray application until death, assessed up to 48 months or lost follow-up, whichever came first
  % of patients who die after Hemospray® application

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study database will be available for other researches. The study protocol is already available at AEG-RedCap platform. STROBE guidelines will be followed.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: July 2018- December 2019
Access Criteria: Accredited researcher or institution. Contact Principal Investigator by email